CLINICAL TRIAL: NCT07399977
Title: A Nonrandomized Trial Using DNA Liquid Biopsies to Guide Anticoagulation For Patients With Cancer-Associated Thromboembolism
Brief Title: Using a Blood Test and Software Tool to Guide Treatment for Venous Thromboembolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-095
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis
Keywords: Venous Thromboembolism; Deep Venous Thrombosis; 25-095; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- High risk for recurrent Venous Thromboembolism/VTE (Experimental): Participants with a ≤5% chance of Venous Thromboembolism/VTE according to the model will be designated "low risk" for the purposes of the study; all other participants will be considered "high risk.
  Interventions: Diagnostic Test: MSK-ACCESS; Diagnostic Test: ctDNA/VTE Risk Score:
- Low-risk for recurrent Venous Thromboembolism/VTE (Experimental): Participants with a ≤5% chance of Venous Thromboembolism/VTE according to the model will be designated "low risk" for the purposes of the study; all other participants will be considered "high risk.
  Interventions: Diagnostic Test: MSK-ACCESS; Diagnostic Test: ctDNA/VTE Risk Score:

INTERVENTIONS:
Diagnostic Test: MSK-ACCESS — MSK-ACCESS is a ctDNA sequencing assay
Diagnostic Test: ctDNA/VTE Risk Score: — Machine learning Venous Thromboembolism/VTE risk score mode

SUMMARY:
The purpose of this study is to find out whether a software tool, ctDNA/VTE (Venous Thromboembolism) risk score model, is an effective way to predict the likelihood of VTE coming back in people who have received anticoagulant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 with a history of cancer-associated VTE (objectively confirmed symptomatic or incidental/unsuspected proximal lower-limb DVT, symptomatic pulmonary embolism [PE] or incidental PE in a segmental or more proximal pulmonary artery) and completion of between 3 and 12 months of anticoagulation with a therapeutic dosing of enoxaparin, dalteparin,rivaroxaban, or apixaban without current VTE-related symptoms (imaging to confirm resolution not required).

Diagnosis of DVT requires evidence of one or more filling defects at compression ultrasonography, venography, CT venography, or MR venography involving at least the popliteal or more proximal veins.

Diagnosis of PE requires an intraluminal filling defect in segmental or more proximal arteries.

* Diagnosis of one of the following solid tumors in either advanced (i.e. unresectable) stage or receiving systemic anticancer treatment within six weeks of enrollment (maintenance therapy included):

  * breast cancer regardless of cytotoxic-chemotherapy status
  * hepatobiliary cancer regardless of cytotoxic-chemotherapy status
  * prostate cancer regardless of cytotoxic-chemotherapy status
  * non-small cell lung cancer with cytotoxic-chemotherapy received within 30 days
  * pancreatic cancer with cytotoxic-chemotherapy received within 30 days
  * bladder cancer with cytotoxic-chemotherapy received within 30 days
* Signed and dated informed consent by study participant/Legally Authorized Representative (LAR).

Exclusion Criteria:

* Contraindication to ongoing anticoagulation
* Contraindication to discontinuation of anticoagulation (examples include but not limited to: known antiphospholipid syndrome or factor V leiden, active arterial thrombus, catheter-associated thrombus, on anticoagulation for atrial fibrillation or other non-oncologic reasons)
* History of major bleeding in the last six months (major bleeding defined as fatal bleeding, and/or symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome; bleeding that necessitates acute surgical intervention; bleeding causing a fall in hemoglobin levels of 1.24 mmol/L (2 g/dL or greater) or more; or bleeding leading to a transfusion of 2 U or more of whole blood or red cells).
* Known diagnosis of disseminated intravascular coagulation (DIC)
* Suspicion for tumor thrombus on the imaging leading to original diagnosis of VTE
* Enrolled in hospice care
* Currently has inferior vena cava (IVC) filter
* Diagnosis of an active hematologic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2030-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of recurrent Venous Thromboembolism/VTE | 6 months
  Evaluate the cumulative incidence of recurrent Venous Thromboembolism/VTE at 6 months following discontinuation of anticoagulation in participants with low risk DNA liquid biopsy-based model.

CONTACTS AND LOCATIONS:
Overall Officials: Justine Jee, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (7):
  - Memorial Sloan Kettering Cancer Center Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York
- Royal North Shore Hospital, Australia, Sydney, Australia

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org